CLINICAL TRIAL: NCT02873273
Title: A Pilot Study of a Dexamethasone Implant System in Humans
Brief Title: Study of a Steroid Delivery System for Pain Relief Treatment in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Figgie (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor-Investigator, Mark Figgie, Chief of the Surgical Arthritis Service, Hospital for Special Surgery, New York
Organization: Hospital for Special Surgery, New York (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-523
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone delivery system (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Sustained delivery system containing 5.0 mg of dexamethasone programmed to release an estimated 10 μg per day

SUMMARY:
The purpose of this study is to determine whether a longer duration, controlled, sustained release dexamethasone delivery system would be more effective in helping patients with osteoarthritis reduce their pain, remain functional, and delay their need for knee replacement.

DETAILED DESCRIPTION:
The objectives of the study are to assess the dexamethasone delivery system for:

* Safety and tolerability
* Efficacy

Formal statistical analysis to compare treatment groups will not be performed due to the small number of participants in this pilot study. Summary statistics will be assessed using the short form of the knee injury and osteoarthritis outcome score (KOOS JR) surveys and questionnaires to assess pain intensity, pain medication consumption and wound assessment.

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥ 40 years of age at time of consent
* Diagnosis of unilateral or bilateral knee osteoarthritis for at least 6 months prior to screening with confirmation of osteoarthritis according to the American College of Rheumatology Criteria for Classification of Idiopathic Osteoarthritis of the Knee (clinical and radiological) based on an X-ray performed within 6 months prior to screening or during the screening period
* Kellgren - Lawrence grade ≥2 on weight bearing anteroposterior femorotibial radiograph performed within 6 months prior to or during screening period
* Mean score of ≥ 5 and ≤ 10 on the 24 hour average pain score (0 - 10 Numeric Rating System) during the screening period
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Willingness to stop all pain medications except acetaminophen and paracetamol 14 days prior to implantation

Exclusion Criteria:

* Fibromyalgia, chronic pain syndrome, or other concurrent medical or arthritic conditions which could interfere with the evaluation of the index knee
* History of inflammatory arthritis including rheumatoid arthritis, juvenile inflammatory arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, reactive arthritis
* Hemophilia
* Achondroplasia
* History of infection in the index joint
* Intra-articular corticosteroid (investigational or marketed) in any joint within three months of screening
* Intra-articular hyaluronic acid (investigational or marketed) in the index knee within three months of screening
* Oral, inhaled, and intranasal corticosteroids (investigational or marketed) within one month of screening
* Prior arthroscopic or open surgery of the index knee within 12 months of screening
* Planned / anticipated surgery of the index knee during the study period
* Active or history of malignancy within the last five years, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ
* Insulin dependent diabetes
* History of or active Cushing's syndrome
* Skin breakdown at index knee where procedure would take place
* Women of child-bearing potential
* Case history related to motor vehicle accident or workers compensation
* Presence of hardware in the index knee (e.g. screws, plates)
* Immunocompromised patients (TB, HIV, etc.)
* Allergic reactions to acetaminophen and paracetamol

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Through 24 weeks
Change from baseline in weekly mean of the pain intensity score | Weeks 12, 24
  Using a numeric rating scale for pain with a scale of 0 (no pain) to 10 (worst pain imaginable) at rest, during activity, and at night

SECONDARY OUTCOMES:
Change from baseline in weekly mean of the pain intensity score | Weekly through 24 weeks
  Using a numeric rating scale for pain with a scale of 0 (no pain) to 10 (worst pain imaginable) at rest, during activity, and at night
Time of onset of pain relief | Weekly through 24 weeks
Change from baseline in KOOS-JR score (stiffness) | Over 1, 2, 4, 8, 12, 24 weeks post treatment
  Using a response scale of none, mild, moderate, severe, and extreme
Change from baseline in KOOS-JR score (pain) | Over 1, 2, 4, 8, 12, 24 weeks post treatment
  Using a response scale of none, mild, moderate, severe, and extreme
Change from baseline in KOOS-JR score (function) | Over 1, 2, 4, 8, 12, 24 weeks post treatment
  Using a response scale of none, mild, moderate, severe, and extreme
Change in patient's global impression of scores assessed via office visits | Weeks 4, 12, 24
  Using a numeric rating scale for pain with a scale of 0 (no pain) to 10 (worst pain imaginable)
Change in clinical observer's global impression of scores assessed via office visits | Weeks 4, 12, 24
  Using a numeric rating scale for pain with a scale of 0 (no pain) to 10 (worst pain imaginable)
Percent of responders (defined as patients with high improvement in pain or function) according to OMERACT-OARSI criteria | Weeks 1, 2, 4, 8, 12, 24
Average weekly consumption of rescue medications | Through 24 weeks
Average total consumption of rescue medications | Through 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Figgie, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No